CLINICAL TRIAL: NCT06501547
Title: Association of Leucocyte Telomere Length With Clinical Examination and Dermoscopic Photoaging Scale (DPAS) Score in Skin Aging: a Pilot Study
Brief Title: Association of Leucocyte Telomere Length With DPAS Score in Skin Aging
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dr.dr.Irma Bernadette, SpKK (K) (Other)
Collaborators: Indonesia Medical Education and Research Institute (Other)
Responsible Party: Sponsor-Investigator, Dr.dr.Irma Bernadette, SpKK (K), Prof. Dr. dr. Irma Bernadette S. Sitohang, Sp.KK (K), Indonesia University
Organization: Indonesia University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: tes
Record Dates: First submitted 2024-06-02; First posted 2024-07-15 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Aging; Skin Laxity
Keywords: Dermoscopy; Dermoscopic photoaging scale (DPAS); Glogau scale; Leucocyte telomere length (LTL); Photoaging; Skin aging; Telomere; Ultraviolet (UV)
MeSH Terms: conditions — Cutis Laxa

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- lifestyle counseling (Experimental): patient will be asked about the mean of sun exposure per week
  Interventions: Genetic: Leucocyte Telomere Length from blood draw
- Clinical examination (Experimental): patients's face were assessed by the doctor by using Glogau scale and the doctor will perform dermoscopic tes to assess dermoscopic photoaging scale (DPAS) score to obtain the score of skin aging
  Interventions: Genetic: Leucocyte Telomere Length from blood draw

INTERVENTIONS:
Genetic: Leucocyte Telomere Length from blood draw — blood draw, PCR method to see leucocyte telomere length

SUMMARY:
The goal is to know the profile of photoaging based on clinical examination, Dermoscopic Photoaging Scale and leucocyte telomere length

The main questions of Research are:

* what is the profile of photoaging based on clinical examination results in skin aging
* what is the profile of photoaging based on DPAS Score in skin aging
* what is the profile of leucocyte telomere length in skin aging

Participants are female and male with the age of 29-31 years old and 59-61 years old. They will be examined by dermatovenereologist and will be photographed in 5 positions, they will get dermocopy on forehead, right cheek , left cheek, and chin, and their blood will be drawn about 10 mL in order to get the profile of leucocyte telomere length

DETAILED DESCRIPTION:
Skin aging is a process of deterioration in the physiological structure and function of the skin that significantly increases in the 4th and 5th decades of life. Skin aging is a combination of physiological and pathological aging. Physiological change cannot be avoided and mandatory for everyone, pathological aging ir extrinsic aging is an abnormal skin condition caused by cigarettes, pollution and ultraviolet (UV). In general, the clinical characteristics of skin aging consist of pigmentation changes, hydration disorders, the appearance of wrinkles and skin tumors. The photoaging assessment was first proposed in 1996 by Dr. Richard Glogau, The Glogau scale assesses photoaging based on clinical assessment grouped into 4 categories, namely types I, II, III, and IV,where each type is graded by the severity of wrinkles, namely from mild, moderate, advanced, and severe. Isik et al. developed an instrument for quantitative skin aging assessment using dermoscopy. This examination is non-invasive and is expected to provide a more objective assessment. There are four facial regions assessed in the DPAS score calculation: forehead, right cheek, left cheek, and chin. The sum of the scores of the four regions is assessed based on 11 parameters, with a maximum final score of 44. Telomeres are repetitive DNA-Protein complexes located at the ends of chromosomes of eukarotic cells, and their function is to maintain chromosome stability during cell division, by protecting chromosomes from degradation and fusion. Many factors affect telomere length, such as body mass index, hormonal therapy, antioxidant intake, chronic diseases, and gender. Research by son et al. found that telomere length shortening was validated to increase the odds of skin aging (OR=0.96, 95% CI: 0.9332-0.99566, P= 0.03) Telomeres are closely linked to cellular aging, especially in dermal cells and telomere shortening in skin fibroblasts may lead to epidermal aging and barrier function defectcs.

ELIGIBILITY:
Inclusion Criteria:

* Female and Male (age 29-31 years old and 59-61 years old
* signs of aging

Exclusion Criteria:

* pregnant or breastfeeding
* have disease or genetic problem

Ages: 29 Years to 61 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
profile of leucocyte telomere length | 1 year
  profile of leucocyte telomere length in skin aging
Profile of skin examination from Glogau scale | 1 year
  Glogau type 1 (mild) is without wrinkles (Age of 28-35 years), type II (moderate) is wrinkles in motion (age of 35-50 years), III (advanced) with wrinkles at rest (age of 50-65 years), type IV (severe) is wrinkles all over the face (age of 60-75)
profile of skin examination with dermoscopic photoaging scale (DPAS) | 1 year
  skin aging is assessed from dermoscopic photoaging scale on dermoscopic images, looking at pigmentary changes, vascular changes, telangiectasis, wrinkles, actinic keratoses, and blackheads. There are four facial regions assessed in the DPAS score calculation, namely the forehead, right cheek, left cheek, and chin. The sum of the scores of the four regions is assessed based on 11 parameters, with a maximum final score of 44.
  The greater the score, the higher marks of skin aging

CONTACTS AND LOCATIONS:
Locations (1):
- Universitas Indonesia, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Yes
provide positive impact for Cipto Mangunkusumo National Hospital and worldwide
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 1 year